CLINICAL TRIAL: NCT06922903
Title: A Multicenter, Open-label, Prospective Phase III Clinical Trial to Evaluate the Diagnostic Efficacy and Safety of INR101 Injection for PET/CT Imaging in Detecting Preoperative Pelvic Lymph Node Metastasis in Patients With Prostate Cancer
Brief Title: Phase III Clinical Trial to Evaluate INR101 Injection for PET/CT Imaging in Patients With Prostate Cancer.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yunhe Pharmaceutical (Tianjin) Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INR101-III-02; CTR20250775 (Other: CDE)
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- INR101 PET/ CT (Experimental): Drug: INR101 7±15% mCi of INR101 will be injected intravenously prior to perform the PET/CT
  Interventions: Drug: INR101

INTERVENTIONS:
Drug: INR101 — INR101

SUMMARY:
A multicenter, open-label, prospective Phase III clinical trial to evaluate INR101 injection for PET/CT imaging in patients with Prostate Cancer

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, single-arm, non-randomized Phase III clinical trial evaluating the diagnostic efficacy and safety of INR101 injection PET/CT imaging in detecting the presence of pelvic lymph node metastasis in participants who are scheduled to undergo radical prostatectomy and pelvic lymph node dissection.

Participants enrolled in clinical trial will receive a single intravenous injection of INR101 injection at a dose of 7 mCi ± 15%, and PET/CT imaging will be performed 80 to 120 minutes after the injection.

The PET/CT images of INR101 injection for each participant will be interpreted independently by two readers blinded to all participant information. When the conclusions of the two readers are inconsistent, a third reader will be added for an adjudication interpretation (the third reader will also be in a blinded during the interpretation process and shall not be aware of the conclusions of the first two readers).

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥18 years old
2. ECOG score of 0 or 1
3. Participants confirmed as prostate adenocarcinoma by histological pathological diagnosis before surgery, and meets the diagnostic criteria for intermediate-risk and above localized prostate cancer in the 2023 CSCO (Chinese Society of Clinical Oncology) guidelines (clinical T stage ≥ T2b; or PSA > 10 ng/mL; or Gleason > 6 score)
4. Intended to undergo radical prostatectomy accompanied by pelvic lymph node dissection
5. Routine blood tests, liver and kidney function, and coagulation function meet the corresponding conditions:

   * Platelet count > 100×10⁹/L.
   * Blood urea nitrogen/urea and serum creatinine ≤ 1.5 x ULN.
   * AST, ALT, and ALP ≤ 2.5 x ULN.
   * Total bilirubin≤ 1.5 x ULN.
   * PT and APTT≤ 1.5 x ULN.
6. Life expectancy of at least 6 months as assessed by investigator
7. Agree to use contraceptive measures from the date of signing the informed consent form to 3 months after medication administration, and avoid sperm donation
8. The participant/legal authorized representative understands the purpose and procedures of the trial and signs the informed consent form

Exclusion Criteria:

1. Participants who are unable to complete the imaging as required
2. Having had ≥ 2 types of malignant tumors within 5 years prior to the first administration, with the exception of fully treated non-metastatic thyroid cancer, basal cell carcinoma of the skin, superficial squamous cell carcinoma of the skin, and superficial bladder cancer.
3. Participants who have previously received, are currently receiving, or plan to receive (from the signing of the informed consent form until the acquisition of the pathological sample) androgen deprivation therapy or any anti-tumor therapy such as radiotherapy, chemotherapy, or endocrine therapy during the trial period.
4. Participants in other interventional clinical trials and within 5 half-lives of the investigational medicinal product or participants in other interventional clinical trials before signing the informed consent form; or participants in clinical trials of radioactive therapeutic drugs before signing the informed consent form and the time from the drug withdrawal to the signing date of the informed consent form is less than 3 months.
5. Have received intravenous iodine contrast agent within 24 hours prior to the administration of INR101, or have received any high-density oral contrast agent within 5 days (except for those who, as judged by the investigator, have no residual contrast agent in the intestines; oral water-soluble contrast agents are acceptable).
6. Participants with a history of salivary gland diseases or Paget's disease
7. Participants with hip joint prostheses
8. Known allergy to the active ingredients of INR101 or its components
9. Serum virology examination, including positive treponema pallidum antibody, positive HIV antibody, positive hepatitis C antibody with positive hepatitis C virus ribonucleic acid (HCV RNA), or active hepatitis B (for those with positive hepatitis B surface antigen, hepatitis B virus deoxyribonucleic acid (HBV DNA) needs to be detected, and if the HBV DNA is positive). (Note: If the investigator assesses and determines that active hepatitis B is not a contraindication for surgery, the participant may be enrolled in the study.)
10. Investigators judge that there are any medical diseases or other conditions that may affect safety, compliance or may affect the study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
With the pathological diagnosis as the standard of truth, the sensitivity and specificity of INR101 injection PET/CT imaging in detecting pelvic lymph node metastasis at the participant level | 30 days after administration
  The sensitivity and specificity of the participant-level will be determined of INR101 injection PET/CT imaging for detection of lesion, confirming against histopathology

SECONDARY OUTCOMES:
With pathological diagnosis as the standard of truth, other diagnostic efficacies of INR101 injection PET/CT imaging in detecting pelvic lymph node metastasis at the participant level, including positive predictive value, negative predictive value and ac | 30 days after administration
  The positive predictive value, negative predictive value and accuracy of the participant -level will be determined of INR101 injection PET/CT imaging for detection of lesion, confirming against histopathology
Compared with conventional imaging examinations, evaluate the difference in the detection rate of distant metastatic lesions (lymph nodes outside the pelvis, viscera/soft tissues and bones) by INR101 injection PET/CT imaging | 30 days after administration
  The detection rate of distant metastatic lesions (lymph nodes outside the pelvis, viscera/soft tissues and bones) will be determined of INR101 injection PET/CT imaging for detection of lesion, comparing with conventional imaging
Assess the consistency of the diagnosis of PET/CT images intra- and inter-reader | 30 days after administration
  The intra- and inter-reader performance will be evaluated by adjudication rate and accept rate
Evaluate the safety and tolerability, including adverse events (AE)/serious adverse events (SAE), vital signs, physical examinations, laboratory tests and 12-lead electrocardiograms | 7 days after administration
  Adverse events will be determined through clinical assessment and categorized by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hongcheng Shi, Principal Investigator — Fudan University; Jianming Guo, Principal Investigator — Fudan University
Locations (32):
- China (32):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No